CLINICAL TRIAL: NCT06395948
Title: A Two-part, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of APG777 in Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study Evaluating APG777 in Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Apogee Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APG777-201
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; APG777; Safety; Efficacy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor's study staff will also be blinded in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Induction Period: APG777 (Experimental): Participants will receive APG777 per protocol defined dosing regimen
  Interventions: Drug: APG777
- Part A: Induction Period: Placebo (Placebo Comparator): Participants will receive matching Placebo injections per protocol defined dosing regimen
  Interventions: Drug: Placebo
- Part A: Maintenance Period: APG777 (Experimental): Participants will receive 1 of 2 maintenance regimens of APG777 per protocol defined dosing regimen
  Interventions: Drug: APG777
- Part B: Induction Period: APG777 (Experimental): Participants will receive APG777 in 1 of 3 regimens per protocol defined dosing regimen
  Interventions: Drug: APG777
- Part B: Induction Period: Placebo (Placebo Comparator): Participants will receive matching placebo injections per protocol defined dosing regimen
  Interventions: Drug: Placebo
- Part B: Maintenance Period: APG777 (Experimental): Participants will receive APG777 per protocol defined dosing regimen
  Interventions: Drug: APG777

INTERVENTIONS:
Drug: APG777 — APG777 subcutaneous injection
  Arms: Part A: Induction Period: APG777; Part A: Maintenance Period: APG777; Part B: Induction Period: APG777; Part B: Maintenance Period: APG777
Drug: Placebo — Matching placebo subcutaneous injection
  Arms: Part A: Induction Period: Placebo; Part B: Induction Period: Placebo

SUMMARY:
This is a two-part study that will evaluate the safety and efficacy of APG777 in participants with moderate-to-severe Atopic Dermatitis (AD). Part A (Proof-of-concept) and Part B (Dose-regimen Finding) will evaluate the safety and efficacy of various induction and maintenance dose regimens of APG777 compared to placebo. The study duration for any individual participant will be up to 106 weeks which includes: screening, induction, maintenance, and post-treatment follow-up periods. Participants randomized in Part A are not permitted to participate in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of AD that has been present for >=1 year prior to the Screening visit
* Moderate-to-severe AD at Screening and Baseline visits
* History of inadequate response to treatment with topical medications, or medical determination that topical therapies are inadvisable
* Applied a stable dose of non-medicated over-the-counter emollient/moisturizer of their choice on their skin for >=14 days prior to Baseline visit and agrees to continue using the same moisturizer throughout the study except the day of the study visits.
* Have completed itch questionnaires in the electronic diary for >=4 of 7 days prior to Baseline visit

Exclusion Criteria:

* Participation in a prior study with APG777.
* Prior treatment with protocol-specified monoclonal antibodies (mAbs)
* Has used any AD-related topical medications within 7 days prior to Baseline visit.
* Has used systemic treatments (other than biologics) and/or phototherapies and/or laser therapy that could affect AD within 4 weeks prior to Baseline visit

Note: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Part A: Percent Change From Baseline in Eczema Area and Severity Index (EASI) | Baseline and at Week 16
Part B: Proportion of participants who achieve EASI 75 at Week 16 | At Week 16

SECONDARY OUTCOMES:
Part A and B: Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 106 Weeks
Part A and B: Change from Baseline in EASI | Baseline, through Week 16 and at Week 52
Part A and B: Percent Change from Baseline in EASI | Baseline through Week 16 and at Week 52
Part A and B: Proportion of Participants Achieving EASI 50, 75, 90, and 100 Score | Baseline through Week 16 and at Week 52
Part A and B: Proportion of Participants Achieving a Validated Investigator Global Assessment (vIGA-AD) Score of 0 (clear) or 1 (almost clear) and a >= 2-Point Reduction | Baseline through Week 16 and at Week 52
Part A and B: Change from Baseline in Body Surface Area (BSA) Involvement | Baseline through Week 16 and at Week 52
Part A and B: Proportion of Participants Achieving a >= 4 Point Improvement in the Weekly Mean of the Daily Itch Numeric Rating Scale (I-NRS) | Baseline through Week 16 and at Week 52
Part A and B: Percent Change from Baseline in the Weekly Mean of the Daily I-NRS | Baseline through Week 16 and at Week 52
Part A and B: Serum Concentrations of APG777 Over Time | Up to 106 Weeks
Part A and B: Predose Serum Concentrations of APG777 (Ctrough) | Up to 106 Weeks
Part A and B: Maximum concentration (Cmax) of APG777 | Up to 106 Weeks
Part A and B: Time to reach Cmax (tmax) | Up to 106 Weeks
Part A and B: Area Under the Concentration-Time Curve (AUC) from Time 0 to Time t (AUC0-t) in the Induction Period | Baseline to 16 Weeks
Part A and B: AUC Over the Dosing Interval (AUC0-tau) in the Maintenance Period | 16 Weeks to 52 Weeks

CONTACTS AND LOCATIONS:
Locations (82):
- United States (28):
  - Investigational Site, Fountain Valley, California
  - Investigational Site, Los Angeles, California
  - Investigational Site, San Diego, California
  - Investigational Site, New Haven, Connecticut
  - Investigational Site, Coral Gables, Florida
  - Investigational Site, Jacksonville, Florida
  - Investigational Site, Margate, Florida
  - Investigational Site, Douglasville, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Skokie, Illinois
  - Investigational Site, West Lafayette, Indiana
  - Investigational Site, Bowling Green, Kentucky
  - Investigational Site, Rockville, Maryland
  - Investigational Site, Detroit, Michigan
  - Investigational Site, Troy, Michigan
  - Investigational Site, Portsmouth, New Hampshire
  - Investigational Site, New York, New York
  - Investigational Site, Wilmington, North Carolina
  - Investigational Site, Boardman, Ohio
  - Investigational Site, Mason, Ohio
  - Investigational Site, Portland, Oregon
  - Investigational Site, Pittsburgh, Pennsylvania
  - Investigational Site, Charleston, South Carolina
  - Investigational Site, Nashville, Tennessee
  - Investigational Site, Dallas, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site, Norfolk, Virginia
  - Investigational Site, Mill Creek, Washington
- Canada (13):
  - Investigational Site, Calgary, Alberta
  - Investigational Site, Edmonton, Alberta
  - Investigational Site, Vancouver, British Columbia
  - Investigational Site, Winnipeg, Manitoba
  - Investigational Site, Fredericton, New Brunswick
  - Investigational Site, Ajax, Ontario
  - Investigational Site, Markham, Ontario
  - Investigational Site, Mississauga, Ontario
  - Investigational Site, Ottawa, Ontario
  - Investigational Site, Peterborough, Ontario
  - Investigational Site, Toronto, Ontario
  - Investigational Site, Montreal, Quebec
  - Investigational Site, Québec, Quebec
- Investigational Site, Prague, Czechia
- France (3):
  - Investigational Site, Rouen, Normandy
  - Investigational Site, Martigues
  - Investigational Site, Nantes
- Germany (15):
  - Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Investigational Site, Heidelberg, Baden-Wurttemberg
  - Investigational Site, Tübingen, Baden-Wurttemberg
  - Investigational Site, Augsburg, Bavaria
  - Investigational Site, München, Bavaria
  - Investigational Site, Blankenfelde-Mahlow, Brandenburg
  - Investigational Site, Darmstadt, Hesse
  - Investigational Site, Frankfurt am Main, Hesse
  - Investigational Site, Bad Bentheim, Lower Saxony
  - Investigational Site, Münster, North Rhine Westfalia
  - Investigational Site, Dresden, Saxony
  - Investigational Site, Kiel, Schleswig-Holstein
  - Investigational Site, Lübeck, Schleswig-Holstein
  - Investigational Site, Berlin
  - Investigational Site, Hamburg
- Hungary (3):
  - Investigational Site, Debrecen, Hajdú-Bihar
  - Investigational Site, Budapest
  - Investigational Site, Szeged
- Poland (9):
  - Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site, Lublin, Lublin Voivodeship
  - Investigational Site, Warsaw, Masovian Voivodeship
  - Investigational Site, Gdansk, Pomeranian Voivodeship
  - Investigational Site, Katowice, Silesian Voivodeship
  - Investigational Site, Sosnowiec, Silesian Voivodeship
  - Investigational Site, Szczecin, West Pomeranian Voivodeship
  - Investigational Site, Krakow, Woj. Małopolskie
  - Investigational Site, Lodz, Łódź Voivodeship
- Spain (7):
  - Investigational Site, Santiago de Compostela, A Coruña
  - Investigational Site, Badalona, Barcelona
  - Investigational Site, Las Palmas de Gran Canaria, Canary Islands
  - Investigational Site, Alicante
  - Investigational Site, Barcelona
  - Investigational Site, Madrid
  - Investigational Site, Zaragoza
- United Kingdom (3):
  - Investigational Site, Salford, Greater Manchester
  - Investigational Site, Dudley, West Midlands
  - Investigational Site, London

IPD SHARING:
Plan to Share IPD: No